CLINICAL TRIAL: NCT06677398
Title: Three Debriefing Methods in Virtual Patient Simulation: a Randomized Controlled Trial
Brief Title: Three Debriefing Methods in Virtual Patient Simulation
Acronym: Debriefing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Saglik Bilimleri Universitesi Gulhane Tip Fakultesi (Other)
Responsible Party: Principal Investigator, Gül ŞAHİN KARADUMAN, Asst. Prof, Saglik Bilimleri Universitesi Gulhane Tip Fakultesi
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Date: 10.09.2024 No:2024-435
Record Dates: First submitted 2024-11-02; First posted 2024-11-06 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Virtual Patient; Debriefing Method; Nursing Student
Keywords: Debriefing; Feedback; Effectiveness; Patient Simulation; Virtual Systems; Nursing Students

STUDY DESIGN:
Intervention Model Description: Parallel group-randomized trial
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Group A (Experimental): Experimental group that used one of the debriefing methods
  Interventions: Other: Debriefing Method 1
- Group B (Experimental): Experimental group that used one of the debriefing methods
  Interventions: Other: Debriefing Method 2
- Group C (Other): A control group that used none of the debriefing methods
  Interventions: Other: Debriefing Method VP

INTERVENTIONS:
Other: Debriefing Method 1 — The researchers used a debriefing method that they chose after a virtual simulation
  Arms: Group A
Other: Debriefing Method VP — The researchers used the debriefing method that virtual patient simulator presents
  Arms: Group C
Other: Debriefing Method 2 — The researchers used a debriefing method that they chose after a virtual simulation
  Arms: Group B

SUMMARY:
In simulation-based training, the debriefing session is considered a cornerstone of learning. Therefore, this study aims to compare two different methods of debriefing sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being 4th grade nursing student at a nursing faculty

Exclusion Criteria:

* Not having participated in simulation before and not having practiced with a virtual patient.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-01-29 (Actual); Study Completion 2025-01-29 (Actual)

PRIMARY OUTCOMES:
Hypothesis 1 | 1 week
  There is a difference in the Simulation Effectiveness Tool scores between students using debriefing methods.
Hypothesis 2 | 1 week
  There is a difference in the Debriefing Experience Scale scores between students using debriefing methods.
Hypothesis 3 | 1 week
  There is a difference in The Student Satisfaction and Self-confidence scores between students using debriefing methods.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Health Sciences Turkey, Gulhane Faculty of Nursing, Ankara, Etlik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Researchers believe that it is important to share the data of the study with other researchers following the completion of the data.

REFERENCES:
- [Background] Dreifuerst, K.T., 2015. Getting started with debriefing for meaningful learning. Clin Simul Nurs 11, 268-275. https://doi.org/10.1016/j.ecns.2015.01.005
- [Background] Decker, S., Alinier, G., Crawford, S.B., Gordon, R.M., Jenkins, D., Wilson, C., 2021. Healthcare Simulation Standards of Best PracticeTM The Debriefing Process. Clin Simul Nurs 58, 27-32. https://doi.org/10.1016/j.ecns.2021.08.011
- [Background] Cheng A, Kessler D, Mackinnon R, Chang TP, Nadkarni VM, Hunt EA, Duval-Arnould J, Lin Y, Cook DA, Pusic M, Hui J, Moher D, Egger M, Auerbach M; International Network for Simulation-based Pediatric Innovation, Research, and Education (INSPIRE) Reporting Guidelines Investigators. Reporting guidelines for health care simulation research: extensions to the CONSORT and STROBE statements. Adv Simul (Lond). 2016 Jul 25;1:25. doi: 10.1186/s41077-016-0025-y. eCollection 2016. PMID 29449994
- See also: Power — https://e-picos.com/apps/power/tisg_c
- See also: Randomly Assign Persons to Groups — https://e-picos.com/apps/calculation/rapg